CLINICAL TRIAL: NCT03960905
Title: A Study the Population Pharmacokinetics of Children Receiving the Anti-infective Drugs for Treatment of Infectious Disease in Central Nervous System
Brief Title: A Study the Population Pharmacokinetics of Children of Infectious Disease in Central Nervous System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wei Zhao (Other)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Wei Zhao, Professor; Head of department of clinical pharmacy and pharmacology, Shandong University
Organization: Shandong University (Other)
Other Study IDs: 2019-CNSI-001
Record Dates: First submitted 2019-04-27; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Central Nervous System Infection
MeSH Terms: conditions — Central Nervous System Infections | interventions — Cefepime; Ceftazidime; Meropenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma and hemocyte
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with the usage of anti-infective drugs: in conformity with the clinical practice
  Interventions: Other: Children with the usage of anti-infective drugs

INTERVENTIONS:
Other: Children with the usage of anti-infective drugs — According to the models of population pharmacokinetics,the investigators and want to correlate use of antibiotics with treatment effectiveness and safety in children.
  Other Names: Cefepime (Maxipime®); ceftazidime; meropenem (Mepem®)

SUMMARY:
The investigators aim to study the population pharmacokinetics of children receiving the anti-infective drugs for treatment of infectious disease in central nervous system.

DETAILED DESCRIPTION:
The investigators aim to study the population pharmacokinetics of children receiving the anti-infective drugs for treatment of infectious disease in central nervous system.In this study, the investigators will detect drug concentration in plasma by using residual blood samples of blood gas analysis and other clinical tests and employ computers for constructing population pharmacokinetic models.

ELIGIBILITY:
Inclusion Criteria:

* Children (29 days-18 years old) with anti-infective therapy against infectious disease in central nervous system.
* Clinical symptoms: acute onset, fever (axillary temperature 38 ℃ or higher), headache, altered level of consciousness, vomiting, irritability, sleepiness, low muscle tone, seizures, before the fontanelle full or uplift, positive meningeal stimulation;
* Aboratory examination: CSF appearance change, CSF routine WBC >100 per ml, CSF routine WBC 10-100 per ml, glucose <40mg/dl, protein >100mg/dl), positive detection of etiology (bacterial culture, antigen detection, gram staining).

Exclusion Criteria:

* autoimmune encephalitis;
* central nervous system infection complicated with tumor;
* allergic to carbapenems or glycopeptide antibiotics;
* other cases not suitable for enrollment (small sample size, incomplete clinical data, etc.).

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with infections of center nurous system therapies.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | up to 4 weeks
  Cmax is a term used in pharmacokinetics refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose.

SECONDARY OUTCOMES:
time to achieve maximum concentration (Tmax) | up to 4 weeks
  Tmax is the term used in pharmacokinetics to describe the time at which the Cmax is observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Beijing Children's Hospital, Capital Medical University, National Center for Children's Health, Beijing, Beijing Municipality, China